CLINICAL TRIAL: NCT05643248
Title: A Single Ascending Dose Pilot Study to Assess the Safety, Tolerability and Pharmacokinetics of NEX-20A Given as a Subcutaneous Prolonged-release Injection to Healthy Male Subjects
Brief Title: To Assess Safety, Tolerability and PK of NEX-20A, a Subcutaneous Prolonged-release Injection to Healthy Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanexa AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEX-20-01
Record Dates: First submitted 2022-11-21; First posted 2022-12-08 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): The planned doses are 15 mg for the sentinel subject in cohort 1 and 35 mg for the remaining 2 subjects in cohort 1
  Interventions: Drug: NEX-20A
- Cohort 2 (Experimental): The planned dose for all 3 subjects in cohort 2 is 70 mg.
  Interventions: Drug: NEX-20A
- Cohort 3 (Experimental): The planned dose for all 3 subjects in the optional cohort 3 is 100 mg.
  Interventions: Drug: NEX-20A

INTERVENTIONS:
Drug: NEX-20A — Subcutaneous prolonged-release injection

SUMMARY:
This is a single-centre, single ascending dose (SAD) pilot study designed to evaluate the safety, tolerability, including local tolerability, and pharmacokinetics (PK) of NEX-20A (lenalidomide) after the administration of a single subcutaneous prolonged-release injection to healthy male volunteers

DETAILED DESCRIPTION:
NEX-20A will be administered in sequential cohorts, 2 standard cohorts and an optional third cohort, each comprising 3 subjects. Subjects will be dosed in a sentinel fashion, and all available safety and tolerability data up until and including 10 days for the sentinel subjects must have been evaluated by the iSRC before dosing the remaining 2 subjects in each cohort.Once safety, tolerability and PK data of the last subject in each cohort has been collected, and interim data analysis has been conducted, there must be at least 1 week between dose escalations.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male subject aged 18 to 65 years, inclusive.
3. Clinically normal medical/surgical history, physical findings, vital signs, 12-lead electrocardiograms (ECGs) and safety laboratory values at the time of screening, as judged by the Investigator.
4. Prospective (male) subjects who are sexually active with female partners must agree to use condoms as well as one of the following highly effective (failure rate <1%) methods of contraception with their partner(s) from 14 days prior to the time of NEX-20A administration until 90 days after the follow-up/end-of-study visit (Visit 14).

   * Previous male sterilization, defined as vasectomy conducted at least 6 months prior to screening with appropriate post-vasectomy documentation of the absence of sperm cells in the ejaculate.
   * Previous female sterilization, defined as tubal ligation or permanent bilateral occlusion of fallopian tubes.
   * Oral (except low-dose gestagen [lynestrenol and norethisterone]), injectable or implanted hormonal contraceptive associated with the inhibition of ovulation.
   * Intrauterine device (IUD).
   * Intrauterine hormone-releasing system (IUS), e.g., progestin-releasing coil

Exclusion Criteria:

1. Body weight outside body mass index 18-30 kg/m2
2. Subjects who intend to father a child during the course of the study, i.e., from screening to the final pregnancy check at Visit 15, or whose female partner is pregnant or currently breastfeeding.
3. Regular smoking or use of nicotine products within the past 6 months prior to screening.

   Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than 3 times/week before the screening visit will be allowed.
4. Any intake of alcohol within the previous 24 hours of screening or subsequent study visits, according to alcohol urine tests.
5. Any positive screen for drugs of abuse at screening or subsequent study visits.
6. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV), according to diagnostic tests.
7. Any use of prescription medication within the previous 14 days of the administration of NEX-20A, at the discretion of the Investigator.
8. Any use of over the counter (non-prescription) medication within the previous 48 hours of the administration of NEX-20A, at the discretion of the Investigator, except occasional intake of paracetamol (maximum 2000 mg/day), as well as nasal decongestants without cortisone, antihistamine or anticholinergics.
9. Regular use of any herbal remedies, vitamins, minerals, and other food supplements, at the discretion of the Investigator, within the previous 14 days of the administration of NEX-20A.
10. Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
11. Dermatological conditions, tattoos or large scars on the abdomen, thigh or upper arm which, in the opinion of the Investigator, may limit the evaluation of local tolerability.
12. History of or current thromboembolic disease, including but not limited to deep vein thrombosis (DVT) and other venous thromboembolisms, untreated hypertension and/or untreated hyperlipidaemia, as judged by the Investigator.
13. Family history of thromboembolic disease, specifically first-degree relative with history of or current thromboembolic disease (see exclusion criterion 12), as judged by the Investigator.
14. History of or current hematologic disorder, including but not limited to thrombocytopenia and/or neutropenia, as judged by the Investigator.
15. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to lenalidomide or drugs with a similar chemical structure or class or to any other ingredient of the formulation/vehicle.
16. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
17. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks prior to the treatment visit (Visit 2).
18. Any planned major surgery within the duration of the study.
19. After 10 minutes supine rest at the time of screening, any vital signs outside the following ranges:

    * Systolic blood pressure: <90 or >140 mmHg, or
    * Diastolic blood pressure <50 or >90 mmHg, or
    * Pulse <40 or >90 bpm
20. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
21. Bilirubin >25 µmol/L, alanine aminotransferase (ALT) >1.1 µkat/L, and/or aspartate aminotransferase (AST) >0.75 µkat/L at the time of screening (all values 1x upper limit of normal [ULN]).
22. Estimated glomerular filtration rate (eGFR) <80 mL/min/1.73 m2 (determined from plasma creatinine by the revised Lund-Malmö GFR estimating equation) at the time of screening.
23. Haemoglobin <130 g/L, absolute neutrophil count (ANC) <1.3x109/L, and/or platelet count <150x109/L at the time of screening.
24. History of or current alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
25. History of or current drug abuse, as judged by the Investigator.
26. History of or current use of anabolic steroids, as judged by the Investigator.
27. Participation in any other clinical study and/or treatment with another investigational drug within 90 days of the treatment visit (Visit 2).
28. Plasma donation within 1 month of screening or blood donation (or corresponding blood loss) during the last 90 days prior to screening.
29. Lack of suitability for participation in the study, for any reason, in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Number of subjects with a clinical significant change from baseline in the systolic blood pressure at 36 days | From first dose until day 36
  Measured in mmHg after 10 minutes supine rest. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the diastolic blood pressure at 36 days | From first dose until day 36
  Measured in mmHg after 10 minutes supine rest. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter PQ/PR at 36 days | From first dose until day 36
  Measured in ms in supine position after 10 minutes of rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter QRS at 36 days | From first dose until day 36
  Measured in ms in supine position after 10 minutes of rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter QT at 36 days | From first dose until day 36
  Measured in ms in supine position after 10 minutes of rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter QTcF at 36 days | From first dose until day 36
  Measured in ms in supine position after 10 minutes of rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the haematology blood parameters measurements at 36 days | From first dose until day 36
  Blood samples for the analysis of haematology will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the clinical chemistry blood laboratory measurements at 36 days | From first dose until day 36
  Blood samples for the analysis of clinical chemistry parameters will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the coagulation parameters blood laboratory measurements at 36 days | From first dose until day 36
  Blood samples for the analysis of clinical coagulation parameters will be collected through venpuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the head at 36 days | From first dose until day 36
  Physical examination including assessment of the head. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of eyes at 36 days | From first dose until day 36
  Physical examination including assessment of the eyes. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the ears at 36 days | From first dose until day 36
  Physical examination including assessment of the ears.Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the nose at 36 days | From first dose until day 36
  Physical examination including assessment of the nose.Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the throat at 36 days | From first dose until day 36
  Physical examination including assessment of the throat. .Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the skin at 36 days | From first dose until day 36
  Physical examination including assessment of the skin. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the thyroid at 36 days | From first dose until day 36
  Physical examination including assessment of the thyroid. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of neurological status at 36 days | From first dose until day 36
  Physical examination including neurological status. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the lungs at 36 days | From first dose until day 36
  Physical examination of the lungs including percussion, inspection, palpation, and auscultation.Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the cardiovascular status of at 36 days | From first dose until day 36
  Physical examination including inspection, palpation, and auscultation of the heart. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the abdomen at 36 days | From first dose until day 36
  Physical examination including assessments of the abdomen (liver and spleen). Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of lymph nodes at 36 days | From first dose until day 36
  Physical examination including assessments of the lymph nodes. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of extremitets at 36 days | From first dose until day 36
  Physical examination including assessments of the extremitets. Descriptive individual data.
Number of subjects with treatment-related adverse events a assessed by frequency | From first dose until day 36
  Number of events.Descriptive individual data.
Number of subjects with treatment-related adverse events a assessed by seriousness | From first dose until day 36
  Seriousness of adverse events.Descriptive individual data.
Number of subjects with treatment-related adverse events a assessed by intensity | From first dose until day 36
  Intensity of adverse events.Descriptive individual data.
Number of subjects with a clinical significant change from baseline in local tolerability i.e skin reactions assessed by visual inspection. | From first dose until day 36
  Visual inspection. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in local tolerability i.e skin reactions assessed by photography. | From first dose until day 36
  Photography of injection site. Descriptive individual data.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 12 hours post-dose on Day 1, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours, 408 hours, 504 hours, 576 hours, 672 hours, 744 hours, 840 hours
  Measurement of lenalidomid
Time of occurrence of Cmax (Tmax) | pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 12 hours post-dose on Day 1, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours, 408 hours, 504 hours, 576 hours, 672 hours, 744 hours, 840 hours
  Measurement of lenalidomid
Area under the plasma concentration vs. time curve (AUC) from time 0 to 8 hours | pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 12 hours post-dose on Day 1, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours, 408 hours, 504 hours, 576 hours, 672 hours, 744 hours, 840 hours
  Measurement of lenalidomid
AUC from time 0 to 12 hours | pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 12 hours post-dose on Day 1, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours, 408 hours, 504 hours, 576 hours, 672 hours, 744 hours, 840 hours
  Measurement of lenalidomid
AUC from time 0 to 7 days | pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 12 hours post-dose on Day 1, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours, 408 hours, 504 hours, 576 hours, 672 hours, 744 hours, 840 hours
  Measurement of lenalidomid
AUC from time 0 to infinity | pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 12 hours post-dose on Day 1, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours, 408 hours, 504 hours, 576 hours, 672 hours, 744 hours, 840 hours
  Measurement of lenalidomid
Terminal elimination half-life | pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 12 hours post-dose on Day 1, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours, 408 hours, 504 hours, 576 hours, 672 hours, 744 hours, 840 hours
  Measurement of lenalidomid

CONTACTS AND LOCATIONS:
Overall Officials: Hjalmar Flygt, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (1):
- CTC Clinical Research Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No